CLINICAL TRIAL: NCT06101381
Title: CD19-directed CAR-T Cell Therapy for Refractory or Relapsed Acute Lymphoblastic Leukemia or Non-Hodgkin Lymphoma: a Multicenter Phase I/II Trial.
Brief Title: CD19-directed CAR-T Cell Therapy for R/R Acute Leukemia and Lymphoma
Acronym: CARTHEDRALL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Blood Center of Ribeirao Preto (Unknown); Hospital das Clínicas de Ribeirão Preto (Other)
Responsible Party: Principal Investigator, Diego Villa Clé, Medical Coordinator, University of Sao Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEMO-02-CART
Record Dates: First submitted 2023-10-04; First posted 2023-10-26 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Leukemia, Acute Lymphoblastic; Lymphoma, Non-Hodgkin
Keywords: Cell therapy; Chimeric antigen receptor T cell; CAR-T cell; CD19; Lymphoma; Acute Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma | interventions — CTL019 chimeric antigen receptor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CD19-directed CAR-T cell (Experimental): After lymphodepletion, a single intravenous infusion of an academic, locally produced, autologous CD19-directed CAR-T cells will be administered.
  Interventions: Biological: CART-19

INTERVENTIONS:
Biological: CART-19 — The academic CART-19 consists of autologous T lymphocytes transduced with a lentiviral vector to express a second-generation chimeric antigen receptor with a single chain variable fragment (scFv) targeting the CD19 antigen conjugated with 4-1BB co-stimulatory and CD3z signaling domains.

SUMMARY:
The goal of this prospective, multicentric, single-arm, phase I/II clinical trial is to evaluate the safety and efficacy of a novel CD19-directed CAR-T cell locally produced in an academic institution in Brazil in patients with refractory or relapsed acute lymphoblastic leukemia or non-Hodgkin lymphoma.

Participants will receive a single intravenous infusion of an autologous academic anti-CD19 CAR-T cell and will be followed for 5 years.

DETAILED DESCRIPTION:
Eighty-one patients with refractory/relapsed (R/R) B acute lymphoblastic leukemia (B-ALL) or non-Hodgkin lymphoma (B-NHL) will be included in this multicentric, phase I/II clinical trial to evaluate the safety and efficacy of a novel academic CD19-directed CAR-T cell developed in Brazil.

After the inclusion of the patient, lymphocyte apheresis will be performed for lymphocyte collection, followed by activation, transduction with a lentiviral vector, and expansion of produced CAR-T cells.

The patient will be hospitalized and receive lymphodepleting chemotherapy started five days before CAR-T cells infusion, with cyclophosphamide (300 mg/m2/day) and fludarabine (30 mg/m2/day) for three days. On Day 0, CAR-T cells will be intravenously administered over 20-30 minutes. The optimal CAR-T cell dose will be 1,7 to 5,4 x106 cells/kg, for ALL patients, and 0,6 to 6,0 x 108 cells (total dose) for NHL patients, but any dose higher than 0,2 x 106 cells/kg (for patients < 50 Kg) or 0,14 x 106 cells/kg and 0,1 x 108 cells (total dose) (for patients ≥ 50Kg), and lower than the maximal 2,6 x 108 cells (total dose) will be infused, depending on the obtained cellular product. During and after infusion, the patient will be monitored for signs and symptoms of toxicity and will remain hospitalized for at least two weeks. All patients will receive anti-viral and anti-pneumocystis prophylaxis. They will be monitored to evaluate treatment efficacy, and acute and late toxicities for five years after infusion.

ELIGIBILITY:
Inclusion Criteria:

For non-Hodgkin Lymphomas (B-NHL):

* Provision of signed Informed Consent form;
* Age between 18 and 70 years;
* Performance status according to the Eastern Cooperative Oncology Group < 2;
* Relapsed or refractory B-NHL of the following types (confirmed by biopsy):

  * Diffuse large B-cell lymphoma (DLBCL, NOS);
  * High-grade B-cell lymphoma (HGBCL);
  * Diffuse large B-cell lymphoma/high-grade B-cell lymphoma with MYC and BCL-2 rearrangement;
  * Follicular lymphoma (FL) grade 3B; or
  * Transformed follicular lymphoma (tFL)
* Refractory or relapsed to two or more lines of systemic therapy, with at least one scheme containing an anti-CD20 monoclonal antibody and anthracycline, as defined below:

  * Refractoriness: partial response (PR), stable disease (SD), or progressive disease (PD) as the best response to the last treatment, assessed by PET-CT, according to the Lugano criteria and confirmed by a new biopsy.
  * Relapsed disease: disease reappearance after obtaining a complete response to the last treatment, assessed by PET-CT, according to the Lugano criteria and confirmed by a new biopsy.
* Have performed, or be ineligible for, autologous hematopoietic progenitor cell transplantation (ASCT). Ineligibility is defined by:

  * Lack of at least partial response after salvage chemotherapy; or
  * Failure to mobilize and/or collect hematopoietic progenitor cells (HPC), as defined by the investigator.
* Measurable disease, defined as:

  * Nodal lesions >15 mm in the long axis, regardless of the length of the short axis, and/or
  * Extranodal lesions (outside lymph node or nodal mass, but including liver and spleen) >10 mm in long axis, regardless of the length of the short axis.
* Adequate organ function:

Renal function defined as:

* estimated glomerular filtration rate (eGFR) ≥ 40 mL/min/1.73 m2

Hepatic function defined as:

* Alanine Transaminase (ALT) and Aspartate Transaminase (AST) ≤ 2.5 × ULN; and
* Total bilirubin ≤ 1.5 × ULN, except for patients with Gilbert syndrome.

Hematologic Function (regardless of transfusions for 14 days) defined as:

* Absolute neutrophil count (ANC) >500/uL
* Platelets ≥ 50,000/uL
* Hemoglobin >7.0 g/dl

  * In women of childbearing potential, willingness to use effective means of birth control for 1 year after CAR-T cell infusion.
  * In male participants, willingness to use a barrier birth control method for 1 year after CAR-T cell infusion
  * Able to comply with inpatient treatment, outpatient treatment, laboratory monitoring, and required clinic visits for the duration of study participation.

For Acute Lymphoblastic Leukemia (B-ALL):

* Provision of signed Informed Consent form;
* Age ≥ 3 and < 25 years;
* Performance status < 2, according to the Eastern Cooperative Oncology Group for patients ≥ 16 years old, or ≥ 50%, according to the Lansky performance status for patients younger than 16 years old;
* Relapsed or refractory CD19 positive B-ALL, with documentation of CD19 disease expression within 3 months of screening visit.
* Relapsed or refractory disease as defined below;

  * Failure to obtain hematologic complete remission (bone marrow with < 5% lymphoblasts by morphologic assessment) after 2 distinct chemotherapy lines; or
  * Relapsed or refractoriness after at least 1 previous chemotherapy regimen and ineligibility for allogeneic hematopoietic progenitor cell transplantation (HSCT) due to lack of available donor (including alternative donors), comorbidity, have previously undergone or refused HSCT; or
  * Relapsed disease ≥ 6 months after HSCT; or
  * Relapsed or refractoriness after ≥ TKi for Philadelphia-positive B-ALL.
* Bone marrow with ≥ 5% lymphoblasts by morphologic assessment within 30 days from screening
* Adequate organ function:

Renal function defined as:

* Estimated glomerular filtration rate (eGFR) ≥ 40 mL/min/1.73 m2

Hepatic function defined as:

* Alanine Transaminase (ALT) and Aspartate Transaminase (AST) ≤ 5 × ULN; and
* Total bilirubin ≤ 2 × ULN, except for patients with Gilbert syndrome.

  * In women of childbearing potential, willingness to use effective means of birth control for 1 year after CAR-T cell infusion.
  * In male participants, willingness to use a barrier birth control method for 1 year after CAR-T cell infusion
  * Able to comply with outpatient treatment, laboratory monitoring, and required clinic visits for the duration of study participation. duration of the parent study and the long-term follow-up observational study

Exclusion Criteria:

For non-Hodgkin Lymphomas (B-NHL):

* Previous or concurrent cancer distinct from B-NHL within 2 years before screening, except for the following:

  * Curatively treated nonmelanomatous skin cancer;
  * Curatively treated cervical carcinoma in situ;
  * Localized breast cancer treated with curative intent with no evidence of active disease; or
  * Localized prostate cancer undergoing active surveillance or anti-androgenic therapy, without evidence of metastatic disease.
* Syndromes and/or genetic diseases with impact on the hematopoietic system, including Down's syndrome, Fanconi anemia, telomeropathies, Li Fraumeni, Blackfan-Diamond anemia, or congenital immunodeficiencies;
* History of previous CAR-T therapy;
* History of previous solid organ transplantation;
* Active central nervous system (CNS) involvement by disease, detected by image or cytology/immunophenotyping of cerebrospinal fluid (CSF);
* Primary central nervous system lymphoma (PCNSL);
* Primary mediastinal large B cell lymphoma (PMBCL);
* Evidence of uncontrolled systemic infection (viral, bacterial, or fungal) which requires IV antibiotics, within 2 weeks before the screening visit;
* Known HIV infection;
* Known HTLV I and II infection;
* History of previous tuberculosis;
* Positive Chagas disease serology;
* Hepatitis B or hepatitis C testing indicating active/ongoing infection, as defined as:

  * HBV: Patients with positive HBsAg are excluded. Patients with positive anti-HBc and negative HBsAg require hepatitis B PCR evaluation before randomization. Patients who are hepatitis B PCR-positive will be excluded.
  * HCV: Patients with positive hepatitis C antibody may be enrolled with a negative result for hepatitis C RNA before study inclusion. Patients who are hepatitis C RNA-positive will be excluded.
* History of a symptomatic CNS disease (or which required treatment within the past year), such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease;
* Significant cardiovascular disease defined as ≥ grade 3 New York Heart Association functional classification system of heart failure, history of myocardial infarction, uncontrolled or symptomatic arrhythmias, or unstable angina within the past 6 months before the screening;
* Chronic lung disease, with hypoxemia (Oxygen saturation measured by pulse oximetry > 93% on room air), or uncontrolled within 4 weeks before the screening visit
* History of an autoimmune disease (including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis) with end-organ damage or requiring systemic immunosuppression/systemic disease-modifying agents in the 2 years preceding the screening visit;

  * Participants with hypothyroidism receiving a stable dose of thyroid replacement hormone may be eligible.
  * Participants with controlled type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
* History of deep vein thrombosis or pulmonary embolism within 6 months before the screening visit, or need to use systemic anticoagulation at the time of screening for any other reason;
* Major surgery within 4 weeks of the screening visit;
* History or suspicion of hemophagocytic lymphohistiocytosis (HLH);
* Vaccination with a live or attenuated virus vaccine within one month before the screening visit;
* Patients with known hypersensitivity, including anaphylaxis, to any component of the investigational treatment;
* Pregnancy, lactation, or plan to get pregnant during the study or within 12 months after CAR-T cell infusion;
* In women of childbearing potential a negative serologic pregnancy test must be obtained 7 days before CAR-T cell infusion;
* Women of childbearing potential, and all male participants, must be willing to observe barrier and highly effective birth control methods (outlined in the study protocol) for 12 months following CAR-T cell infusion;
* Presence of any other medical condition that in the investigator's opinion may interfere with the safety or effectiveness evaluation of the study;
* Life expectancy less than 12 weeks, by investigator assessment.

For Acute Lymphoblastic Leukemia (B-ALL)::

* Previous or concurrent cancer distinct from B-NHL within 2 years before screening, except for the following:

  * Curatively treated nonmelanomatous skin cancer;
  * Curatively treated cervical carcinoma in situ;
  * Localized breast cancer treated with curative intent with no evidence of active disease; or
  * Localized prostate cancer undergoing active surveillance or anti-androgenic therapy, without evidence of metastatic disease.
* Syndromes and/or genetic diseases with impact on the hematopoietic system, including Down's syndrome, Fanconi anemia, telomeropathies, Li Fraumeni, Blackfan-Diamond anemia, or congenital immunodeficiencies;
* Isolated extramedullary disease;
* Active central nervous system (CNS) involvement by disease (CNS-3 according to NCCN guideline), detected by cytology/immunophenotyping of cerebrospinal fluid (CSF) within 30 days from screening visit.

  * Patients with CNS-1 and CNS-2 within 30 days from screening visit may be enrolled;
* Burkitt's Leukemia/Lymphoma
* Active acute or chronic graft-versus-host disease (GvHD), or controlled with immunosuppressants in the previous 12 weeks before the screening visit;
* Failure to obtain hematologic complete remission (bone marrow with < 5% lymphoblasts by morphologic assessment) after an anti-CD19 antibody-containing treatment (e.g. Blinatumomab);
* History of previous CAR-T therapy;
* History of previous solid organ transplantation;
* Evidence of uncontrolled systemic infection (viral, bacterial, or fungal) which requires IV antibiotics, within 2 weeks before the screening visit;
* Known HIV infection;
* Known HTLV I and II infection;
* History of previous tuberculosis;
* Positive Chagas' disease serology;
* Hepatitis B or hepatitis C testing indicating active/ongoing infection, as defined as:

  * HBV: Patients with positive HBsAg are excluded. Patients with positive anti-HBc and negative HBsAg require hepatitis B PCR evaluation before randomization. Patients who are hepatitis B PCR-positive will be excluded.
  * HCV: Patients with positive hepatitis C antibody may be enrolled with a negative result for hepatitis C RNA before study inclusion. Patients who are hepatitis C RNA-positive will be excluded.
* History of a symptomatic CNS disease (or which required treatment within the past year), such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease;
* Significant cardiovascular disease defined as ≥ grade 3 New York Heart Association functional classification system of heart failure, history of myocardial infarction, uncontrolled or symptomatic arrhythmias, or unstable angina within the past 6 months before the screening;
* Chronic lung disease, with hypoxemia (Oxygen saturation measured by pulse oximetry > 93% on room air), or uncontrolled within 4 weeks before the screening visit
* History of an autoimmune disease (including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis) with end-organ damage or requiring systemic immunosuppression/systemic disease-modifying agents in the 2 years preceding the screening visit;

  * Participants with hypothyroidism receiving a stable dose of thyroid replacement hormone may be eligible.
  * Participants with controlled type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
* History of deep vein thrombosis or pulmonary embolism within 6 months before the screening visit, or need to use systemic anticoagulation at the time of screening for any other reason;
* Major surgery within 4 weeks of the screening visit;
* History or suspicion of hemophagocytic lymphohistiocytosis (HLH);
* Vaccination with a live or attenuated virus vaccine within one month before the screening visit;
* Patients with known hypersensitivity, including anaphylaxis, to any component of the investigational treatment;
* Pregnancy, lactation, or plan to get pregnant during the study or within 12 months after CAR-T cell infusion;
* In women of childbearing potential a negative serologic pregnancy test must be obtained 7 days before CAR-T cell infusion;
* Women of childbearing potential, and all male participants, must be willing to observe barrier and highly effective birth control methods (outlined in the study protocol) for 12 months following CAR-T cell infusion;
* Presence of any other medical condition that in the investigator's opinion may interfere with the safety or effectiveness evaluation of the study;
* Life expectancy less than 12 weeks, by investigator assessment.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Safety: Number of participants who experience early adverse events. | From patient's inclusion until 30 days after CAR-T cell infusion
  To evaluate the occurrence of early adverse events related to the study treatment, from inclusion until 30 days after CAR-T cell infusion.
Safety: Number of participants who experience late adverse events. | From week 5 to week 52
  To evaluate the occurrence of early adverse events related to the study treatment, from week 5 to week 52.

SECONDARY OUTCOMES:
Efficacy: Overall Response Rate (ORR) | Day 30 and day 90 after CAR-T cell infusion
  The combined number of participants achieving Complete Response (CR) or Partial Response (PR) as the best response at day 30 and day 90 after CAR-T cell infusion, determined by the investigators, following Lugano criteria in non-Hodgkin lymphomas; or the combined number of participants achieving Complete Remission (CR) or Complete Remission with Incomplete Hematologic Recovery (CRi) as the best response at day 30 and day 90 after CAR-T cell infusion, determined by the investigators, in Acute Lymphoblastic Leukemia.
Efficacy: Event Free Survival (EFS) | From patient's inclusion until 5 years
  The time between patient's inclusion and relapse, disease progression, or death of any cause.
Efficacy: Relapse Free Survival (RFS) | From patient's inclusion until 5 years
  The duration of response, defined as the time from the first complete or partial response to the date of first documentation of relapse, disease progression, or death of any cause.
Efficacy: Overall Survival (EFS) | From patient's inclusion until 5 years
  The number of participants surviving since patient's inclusion until 5 years

OTHER OUTCOMES:
Exploratory: Number of patientes with CAR-T cell persistence over the time | From CAR-T cell infusion until 5 years
  To evaluate the persistence of infused CAR-T cells in patient's peripheral blood over the time
Exploratory: Replication-competent lentivirus (RCL) | From CAR-T cell infusion until 5 years
  To evaluate the presence of replication-competent lentivirus in patient's peripheral blood, after CAR-T cell infusion, in a cohort of 10 patients.

CONTACTS AND LOCATIONS:
Overall Officials: Diego V Cle, MD, PhD, MBA, Principal Investigator — Ribeirao Preto School of Medicine, University of Sao Paulo
Locations (5):
- Brazil (5):
  - Hospital de Clínicas da UNICAMP, Campinas, São Paulo
  - Ribeirao Preto School of Medicine, University of Sao Paulo, Ribeirão Preto, São Paulo
  - Hospital Sírio-Libanês, São Paulo, São Paulo
  - Hospital das Clinicas de São Paulo, São Paulo, São Paulo
  - A Beneficência Portuguesa de São Paulo, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No